CLINICAL TRIAL: NCT02516605
Title: A Multi-part, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Efficacy of Tropifexor (LJN452) in Patients With Primary Biliary Cholangitis
Brief Title: A Multi-part, Double Blind Study to Assess Safety, Tolerability and Efficacy of Tropifexor (LJN452) in PBC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLJN452X2201; 2015-001590-41 (EudraCT Number)
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-10

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cirrhosis, PBC; Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — tropifexor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LJN452 (Experimental)
  Interventions: Drug: Part 1: LJN452; Drug: Part 2: LJN452 Dose level 1; Drug: Part 2: LJN452 Dose level 2
- Placebo (Placebo Comparator)
  Interventions: Drug: Part 1: Placebo; Drug: Part 2: Placebo

INTERVENTIONS:
Drug: Part 1: LJN452 — LJN452 capsules administered once daily for 28 days
  Other Names: tropifexor
  Arms: LJN452
Drug: Part 1: Placebo — Matching placebo capsules administered once daily for 28 days
  Arms: Placebo
Drug: Part 2: LJN452 Dose level 1 — LJN452 capsules administered once a day for 12 weeks
  Other Names: tropifexor
  Arms: LJN452
Drug: Part 2: Placebo — Matching placebo to LJN452 administered once a day for 12 weeks
  Arms: Placebo
Drug: Part 2: LJN452 Dose level 2 — LJN452
  Other Names: tropifexor
  Arms: LJN452

SUMMARY:
A multi-part study to assess safety, tolerability and efficacy of tropifexor (LJN452) in patients with primary biliary cholangitis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of PBC as demonstrated by the presence of at least 2 of the following 3 diagnostic criteria:

  * History of alkaline phosphatase (ALP) elevated above upper limit of normal (ULN) for at least 6 months
  * Positive antimitochondrial antibodies (AMA) titer or if AMA negative or in low titer (<1:80) PBC specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components (PDC-E2, 2-oxo-glutaric acid dehydrogenase complex))
  * Previous liver biopsy findings consistent with PBC
* At least 1 of the following markers of disease severity:

  * ALP ≥ 1.67 × ULN
  * Total bilirubin > ULN but < 1.5 × ULN
* In addition, patients must meet the following biochemical criteria at enrollment:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 × ULN
  * Total bilirubin ≤ 1.5 × ULN
  * INR ≤ ULN
* Taking UDCA for at least 12 months, or for at least 6 months and has reached maximal response to UDCA with a plateau in alkaline phosphatase, with no changes in dose for ≥ 3 months prior to Day 1.
* Patients must weigh at least 40 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 40 kg/m2. BMI = Body weight (kg) / [Height (m)]2

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception for 30 days before randomization, during dosing and for 30 days following the end of treatment.
* Presence of other concomitant liver diseases.

  * Cirrhosis with complications, including history or presence of:
  * Variceal bleed
  * Uncontrolled ascites
  * Encephalopathy
  * Spontaneous bacterial peritonitis
* Significant hepatic impairment as defined by Child-Pugh classification of B or C, history of liver transplantation, current placement on a liver transplant list or current Model for End Stage Liver Disease (MELD) score ≥15.
* History of conditions that may cause increases in ALP (e.g., Paget's disease).
* Use of investigational drugs, or immunosuppressive drugs at the time of enrollment, or within 5 half-lives, or 30 days of randomization, whichever is longer; or longer if required by local regulations. Use of high dose oral steroids to treat co-morbid conditions (e.g., airways disease) will be allowed but must be properly documented as such in concomitant medications.
* Currently taking obeticholic acid or have taken obeticholic acid within 30 days of randomization
* Previous participation in CLJN452X2201 and received study medication within three months of randomization (or longer if required by local regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (9):
  - Novartis Investigative Site, Rialto, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Manhasset, New York
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Seattle, Washington
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
- Germany (5):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Poland (4):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Mysłowice
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
- United Kingdom (5):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Schramm C, Wedemeyer H, Mason A, Hirschfield GM, Levy C, Kowdley KV, Milkiewicz P, Janczewska E, Malova ES, Sanni J, Koo P, Chen J, Choudhury S, Klickstein LB, Badman MK, Jones D. Farnesoid X receptor agonist tropifexor attenuates cholestasis in a randomised trial in patients with primary biliary cholangitis. JHEP Rep. 2022 Jul 21;4(11):100544. doi: 10.1016/j.jhepr.2022.100544. eCollection 2022 Nov. PMID 36267872
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=322

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study comprised of an escalating multiple dose design in PBC patients with incomplete biochemical response to, but still taking, ursodeoxycholic acid (UDCA).
Groups:
- LJN452 - 0.03 mg qd: Tropifexor 0.03 mg daily for 28 days
- LJN452 - 0.06 mg qd: Tropifexor 0.06 mg daily for 28 days
- LJN452 - 0.09 mg qd: Tropifexor 0.09 mg daily for 28 days
- LJN452 - 0.15 mg qd: Tropifexor 0.15 mg daily for 28 days
- Placebo qd: Tropifexor placebo daily for 28 days
Period: Overall Study
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Started | 11 | 9 | 12 | 8 | 21
Completed | 11 | 9 | 12 | 7 | 20
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all subjects who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd | Total
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.42) | 57.9 (11.21) | 53.6 (7.42) | 57.4 (13.81) | 53.7 (10.19) | 55.7 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 12 | 8 | 21 | 59
  Male | 0 | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 10 | 8 | 12 | 8 | 19 | 57
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Other | 1 | 1 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Serum Gamma-glutamyl Transferase (GGT)
Description: Fold change in serum gamma-glutamyl transferase (GGT) from baseline to Day 28
Time Frame: Baseline to Day 28
Population: The PD analysis set included all subjects with any available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (90% Confidence Interval); unit: fold-change
Groups:
- Pooled Placebo: Placebo data from all cohorts were pooled.
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Pooled Placebo
Number analyzed (Participants) | 10 | 9 | 12 | 8 | 20
fold-change | 0.74 [0.61 to 0.90] | 0.41 [0.33 to 0.50] | 0.28 [0.23 to 0.33] | 0.31 [0.24 to 0.40] | 0.86 [0.75 to 0.99]
Statistical Analysis 1: Comparison: LJN452 - 0.03 mg qd vs Pooled Placebo; Test type: Other; p = 0.293, ANCOVA; adjusted fold change from baseline = 0.86, 90% CI 2-sided [0.68 to 1.09]
Statistical Analysis 2: Comparison: LJN452 - 0.06 mg qd vs Pooled Placebo; Test type: Other; p < 0.001, ANCOVA; adjusted fold change from baseline = 0.47, 90% CI 2-sided [0.37 to 0.60]
Statistical Analysis 3: Comparison: LJN452 - 0.09 mg qd vs Pooled Placebo; Test type: Other; p < .001, ANCOVA; adjusted fold change from baseline = 0.32, 90% CI 2-sided [0.26 to 0.40]
Statistical Analysis 4: Comparison: LJN452 - 0.15 mg qd vs Pooled Placebo; Test type: Other; p < .001, ANCOVA; adjusted fold change from baseline = 0.36, 90% CI 2-sided [0.27 to 0.47]

2. Primary Outcome: Blood Pressure
Description: Vital signs - Systolic Blood pressure
Time Frame: Screening, Baseline, day 1, day 7, day 14, day 21, day 28, day 56, day 84
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21
mm Hg
  Screening | 122.5 (12.21) | 125.8 (11.79) | 129.3 (14.42) | 129.5 (17.42) | 123.0 (15.40)
  Baseline | 124.7 (17.66) | 128.4 (13.83) | 122.0 (18.18) | 132.3 (18.09) | 118.7 (12.76)
  Day 1 | 129.6 (20.48) | 122.4 (20.24) | 119.9 (11.84) | 129.1 (25.12) | 123.0 (21.84)
  Day 7: number analyzed (Participants) | 11 | 9 | 12 | 8 | 20
  Day 7 | 127.2 (20.18) | 123.7 (13.04) | 125.6 (14.22) | 128.0 (26.58) | 120.9 (19.57)
  Day 14: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  Day 14 | 122.4 (16.30) | 124.6 (20.67) | 127.1 (16.45) | 127.3 (12.45) | 118.7 (12.88)
  Day 21: number analyzed (Participants) | 11 | 9 | 12 | 6 | 20
  Day 21 | 121.5 (11.25) | 126.3 (27.65) | 123.9 (13.14) | 124.0 (14.23) | 124.5 (19.8)
  Day 28: number analyzed (Participants) | 11 | 9 | 12 | 5 | 20
  Day 28 | 118.0 (11.22) | 127.1 (28.55) | 121.4 (12.82) | 126.0 (7.71) | 120.1 (22.38)
  Day 56: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  Day 56 | 121.4 (10.76) | 125.4 (18.48) | 121.5 (11.55) | 129.1 (26.45) | 123.8 (19.74)
  Day 84 | 131.3 (16.04) | 124.6 (15.77) | 122.3 (7.70) | 130.4 (25.51) | 123.6 (19.09)

3. Primary Outcome: Pulse Rate
Description: Vital signs
Time Frame: Screening, Baseline, day 1, day 7, day 14, day 21, day 28, day 56, day 84
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21
bpm
  Screening | 68.6 (10.63) | 61.2 (7.05) | 75.3 (8.22) | 72.8 (8.26) | 69.3 (10.69)
  Baseline | 64.3 (7.79) | 64.1 (8.70) | 70.8 (8.63) | 74.4 (5.15) | 66.3 (9.30)
  Day 1 | 67.7 (11.93) | 64.2 (8.07) | 69.7 (7.50) | 74.1 (11.62) | 67.6 (8.35)
  Day 7: number analyzed (Participants) | 11 | 9 | 12 | 8 | 20
  Day 7 | 65.2 (9.98) | 66.8 (11.31) | 70.1 (11.64) | 73.5 (8.33) | 65.2 (8.92)
  Day 14: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  Day 14 | 62.9 (10.03) | 64.8 (8.09) | 70.5 (14.16) | 75.1 (6.74) | 66.1 (9.61)
  Day 21: number analyzed (Participants) | 11 | 9 | 12 | 6 | 20
  Day 21 | 65.5 (8.26) | 65.8 (11.18) | 73.2 (8.43) | 72.5 (6.75) | 67.7 (10.18)
  Day 28: number analyzed (Participants) | 11 | 9 | 12 | 5 | 20
  Day 28 | 65.5 (10.83) | 68.9 (10.60) | 68.5 (9.01) | 67.2 (3.42) | 65.8 (9.29)
  Day 56: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  Day 56 | 66.8 (9.64) | 67.7 (7.53) | 69.7 (8.17) | 69.7 (4.07) | 68.1 (10.11)
  Day 84 | 65.6 (10.24) | 64.0 (9.11) | 70.2 (8.14) | 72.8 (8.12) | 68.1 (9.82)

4. Primary Outcome: Body Temperature
Description: Vital signs
Time Frame: Screening, Baseline, day 1, day 7, day 14, day 21, day 28, day 56, day 84
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21
Celsius
  Screening: number analyzed (Participants) | 11 | 9 | 12 | 8 | 20
  Screening | 36.605 (0.2813) | 36.567 (0.2000) | 36.424 (0.3429) | 36.650 (0.1604) | 36.460 (0.4500)
  baseline | 36.582 (0.2960) | 36.644 (0.2128) | 36.398 (0.3385) | 36.638 (0.1506) | 36.376 (0.5118)
  day 1 | 36.436 (0.3139) | 36.537 (0.3076) | 36.482 (0.2636) | 36.575 (0.1982) | 36.390 (0.4867)
  day 7: number analyzed (Participants) | 11 | 9 | 12 | 8 | 20
  day 7 | 36.582 (0.2040) | 36.533 (0.1323) | 36.258 (0.3965) | 36.600 (0.1195) | 36.345 (0.4639)
  day 14: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  day 14 | 36.516 (0.1793) | 36.444 (0.2007) | 36.291 (0.4109) | 36.500 (0.1826) | 36.310 (0.4576)
  day 21: number analyzed (Participants) | 11 | 9 | 12 | 6 | 20
  day 21 | 36.500 (0.2490) | 36.267 (0.4637) | 36.308 (0.3288) | 36.433 (0.1966) | 36.455 (0.4236)
  day 28: number analyzed (Participants) | 11 | 9 | 12 | 5 | 20
  day 28 | 36.382 (0.2228) | 36.444 (0.2128) | 36.308 (0.3397) | 36.520 (0.2950) | 36.380 (0.4047)
  day 56: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  day 56 | 36.527 (0.2102) | 36.500 (0.2179) | 36.350 (0.4602) | 36.443 (0.3309) | 36.285 (0.4246)
  day 84 | 36.482 (0.2483) | 36.500 (0.1500) | 36.383 (0.2980) | 36.638 (0.1506) | 36.295 (0.4248)

5. Primary Outcome: ECG - Heart Rate
Description: Electrocardiogram (ECG)
Time Frame: Screening, Baseline, day 1, day 28
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21
bpm
  Screening: number analyzed (Participants) | 10 | 9 | 12 | 8 | 21
  Screening | 65.8 (11.32) | 61.8 (9.97) | 67.3 (5.58) | 67.8 (6.54) | 63.4 (9.35)
  Baseline | 60.5 (8.99) | 61.4 (8.75) | 64.6 (7.95) | 67.9 (6.45) | 63.8 (9.41)
  Day 1 | 61.5 (11.16) | 63.4 (11.17) | 63.9 (8.21) | 66.9 (11.97) | 63.5 (7.12)
  Day 28: number analyzed (Participants) | 11 | 9 | 12 | 5 | 20
  Day 28 | 60.5 (11.39) | 65.2 (11.95) | 63.5 (9.95) | 65.8 (4.55) | 60.8 (7.03)

6. Primary Outcome: ECG Intervals - PR Interval
Description: Electrocardiogram (ECG)
Time Frame: Screening, Baseline, day 1, day 28
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21
msec
  Screening: number analyzed (Participants) | 10 | 9 | 12 | 8 | 21
  Screening | 159.2 (27.34) | 158.0 (23.71) | 172.0 (24.12) | 159.9 (17.24) | 162.6 (19.03)
  Baseline | 165.8 (20.81) | 156.2 (18.99) | 175.0 (34.96) | 152.0 (22.21) | 160.3 (19.77)
  Day 1 | 165.5 (21.76) | 162.9 (27.06) | 175.7 (28.29) | 160.0 (20.32) | 161.6 (20.28)
  Day 28: number analyzed (Participants) | 11 | 9 | 12 | 5 | 20
  Day 28 | 164.9 (19.75) | 157.1 (26.70) | 180.4 (31.63) | 155.4 (23.51) | 160.2 (28.70)

7. Primary Outcome: Haemoglobin
Description: Hematology panel for safety laboratory assessments.
Time Frame: Screening, Baseline, day 1, day 7, day 14, day 21, day 28, day 56, day 84
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 11 | 9 | 12 | 8 | 21
g/L
  Screening | 127.9 (9.24) | 125.6 (11.70) | 130.5 (9.73) | 133.9 (12.70) | 132.2 (8.81)
  baseline | 126.5 (8.58) | 127.4 (11.85) | 130.5 (11.90) | 134.6 (13.24) | 131.3 (8.02)
  day 1 | 124.7 (8.21) | 132.9 (10.05) | 127.0 (9.03) | 133.1 (11.37) | 126.8 (7.63)
  day 7: number analyzed (Participants) | 11 | 9 | 12 | 8 | 20
  day 7 | 124.0 (8.23) | 128.8 (16.97) | 132.4 (10.66) | 134.0 (8.75) | 128.6 (9.18)
  day 14: number analyzed (Participants) | 11 | 9 | 12 | 7 | 20
  day 14 | 126.5 (9.83) | 127.3 (12.64) | 128.6 (7.82) | 135.4 (13.50) | 128.7 (10.84)
  day 21: number analyzed (Participants) | 11 | 9 | 12 | 6 | 20
  day 21 | 127.5 (8.32) | 128.0 (13.49) | 130.5 (10.40) | 134.2 (9.91) | 128.8 (10.79)
  day 28: number analyzed (Participants) | 10 | 9 | 12 | 5 | 20
  day 28 | 125.3 (9.18) | 127.1 (14.67) | 129.6 (10.02) | 136.4 (13.50) | 125.7 (9.71)
  day 56: number analyzed (Participants) | 11 | 8 | 12 | 5 | 20
  day 56 | 126.7 (6.96) | 125.8 (11.15) | 128.6 (10.63) | 133.6 (12.00) | 129.3 (11.39)
  day 84 | 126.5 (8.78) | 124.9 (9.75) | 125.9 (11.19) | 131.1 (10.91) | 129.3 (9.24)

8. Secondary Outcome: Plasma PK Parameter - AUC 0-8h
Description: Tropifexor levels were determined in plasma using a validated LC-MS/MS method. AUC0-t=The area under the plasma concentration-time curve from time zero to time 't' where t is a defined time point after administration [mass x time / volume]
Time Frame: Day 1, Day 28
Population: The PK analysis set included all subjects with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd
Number analyzed (Participants) | 9 | 7 | 3 | 4
hr*ng/mL
  Day 1: number analyzed (Participants) | 7 | 3 | 0 | 4
  Day 1 | 4.98 (2.87) | 12.1 (2.68) |  | 24.5 (15.9)
  Day 28: number analyzed (Participants) | 9 | 7 | 3 | 3
  Day 28 | 7.95 (4.21) | 17.6 (5.30) | 23.4 (8.70) | 44.2 (25.8)

9. Secondary Outcome: Plasma PK Parameter - Cmax
Description: Tropifexor levels were determined in plasma using a validated LC-MS/MS method. Cmax=The observed maximum plasma concentration following drug administration [mass /volume]
Time Frame: Day 1, Day 28
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd
Number analyzed (Participants) | 11 | 9 | 12 | 8
ng/mL
  Day 1: number analyzed (Participants) | 10 | 7 | 12 | 8
  Day 1 | 1.04 (0.484) | 1.80 (0.585) | 2.37 (1.56) | 4.84 (2.59)
  Day 28: number analyzed (Participants) | 11 | 9 | 12 | 4
  Day 28 | 1.25 (0.559) | 2.55 (0.946) | 4.30 (2.10) | 6.37 (3.40)

10. Secondary Outcome: Plasma PK Parameter - Tmax
Description: Tropifexor levels were determined in plasma using a validated LC-MS/MS method. Tmax = The time to reach the maximum concentration after drug administration [time]
Time Frame: Day 1, Day 28
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd
Number analyzed (Participants) | 11 | 9 | 12 | 8
hr
  Day 1: number analyzed (Participants) | 10 | 7 | 12 | 8
  Day 1 | 4.12 [2.00 to 8.00] | 4.00 [3.70 to 6.00] | 4.00 [0 to 7.83] | 4.00 [4.00 to 4.18]
  Day 28: number analyzed (Participants) | 11 | 9 | 12 | 4
  Day 28 | 4.08 [2.00 to 8.00] | 4.00 [3.13 to 7.60] | 4.00 [0 to 6.00] | 5.00 [3.03 to 6.00]

11. Secondary Outcome: Changes From Baseline in Total PBC-40 Score
Description: Baseline is defined as the latest available predose value. The PBC-40 is a paper-based, patient-derived, disease-specific health-related quality of life (HRQOL) patient reported outcome (PRO) measure which was developed and validated for use in PBC patients (Jacoby et al 2005). It consists of 40 questions arranged in 6 domains with between 3 and 11 questions in each domain. Each question is scored from 1 to 5 in increasing order of severity. All questions within a domain are summed and all domain totals are summed to obtain a total score. The total score range is between a minimum of 40 and a maximum of 200. Higher scores represent a poorer quality of life. The median difference from baseline in total sum score for each treatment group is presented.
Time Frame: Baseline, Day 28, Day 56, Day 84
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 10 | 9 | 12 | 8 | 20
units on a scale
  Day 28: number analyzed (Participants) | 9 | 9 | 12 | 5 | 18
  Day 28 | 2.0 [-10 to 7] | 1.0 [-14 to 16] | 3.5 [-7 to 13] | -1.0 [-5 to 43] | -2.0 [-23 to 26]
  Day 56: number analyzed (Participants) | 9 | 9 | 12 | 7 | 18
  Day 56 | 3.0 [-7 to 29] | 3.0 [-15 to 23] | -2.5 [-15 to 16] | -3.0 [-28 to 3] | 1.0 [-12 to 30]
  Day 84: number analyzed (Participants) | 9 | 9 | 12 | 8 | 18
  Day 84 | -2.0 [-12 to 13] | -1.0 [-14 to 16] | -3.5 [-38 to 10] | -1.0 [-12 to 5] | 1.5 [-38 to 30]
Statistical Analysis 1: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.898, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 1.0, 90% CI 2-sided [-7.0 to 6.0]
Statistical Analysis 2: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.593, Wilcoxon rank-sum test; Day 56; Median difference from baseline = 2.0, 90% CI 2-sided [-4.0 to 10.0]
Statistical Analysis 3: Comparison: LJN452 - 0.03 mg qd; Test type: Other; p = 0.509, Wilcoxon rank-sum test; Day 84; Median difference from baseline = -3.0, 90% CI 2-sided [-11.0 to 4.0]
Statistical Analysis 4: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.591, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 1.5, 90% CI 2-sided [-5.0 to 7.0]
Statistical Analysis 5: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.702, Wilcoxon rank-sum test; Day 56; Median difference from baseline = -2.0, 90% CI 2-sided [-12.0 to 4.0]
Statistical Analysis 6: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.838, Wilcoxon rank-sum test; Day 84; Median difference from baseline = -1.0, 90% CI 2-sided [-10.0 to 8.0]
Statistical Analysis 7: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.297, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 4.0, 90% CI 2-sided [-3.0 to 8.0]
Statistical Analysis 8: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.236, Wilcoxon rank-sum test; Day 56; Median difference from baseline = -6.0, 90% CI 2-sided [-14.0 to 1.0]
Statistical Analysis 9: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.192, Wilcoxon rank-sum test; Day 84; Median difference from baseline = -6.5, 90% CI 2-sided [-15.0 to 1.0]
Statistical Analysis 10: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.605, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 2.0, 90% CI 2-sided [-2.0 to 9.0]
Statistical Analysis 11: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.037, Wilcoxon rank-sum test; Day 56; Median difference from baseline = -11.0, 90% CI 2-sided [-21.0 to -1.0]
Statistical Analysis 12: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.397, Wilcoxon rank-sum test; Day 84; Median difference from baseline = -3.5, 90% CI 2-sided [-11.0 to 3.0]

12. Secondary Outcome: Change From Baseline in Itch Subdomain of PBC-40 Score
Description: Baseline is defined as the latest available predose value. The PBC-40 is a paper-based, patient-derived, disease-specific health-related quality of life (HRQOL) patient reported outcome (PRO) measure which was developed and validated for use in PBC patients (Jacoby et al 2005). It consists of 40 questions arranged in 6 domains with between 3 and 11 questions in each domain. Each question is scored from 1 to 5 in increasing order of severity. This dataset focuses on the itch subdomain which consists of 3 questions. These 3 questions within the itch subdomain are summed to obtain a total score for the itch subdomain. The total score range is between a minimum of 3 and a maximum of 15. Higher scores represent a poorer quality of life. The median change from baseline in total itch subdomain score in each treatment group is presented.
Time Frame: Baseline, Day 28, Day 56, Day 84
Population: as for outcome 1
Measure: Median (Full Range); unit: UNITS ON A SCALE
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 10 | 9 | 12 | 8 | 20
UNITS ON A SCALE
  Day 28: number analyzed (Participants) | 9 | 9 | 12 | 5 | 18
  Day 28 | 1.0 [-2 to 7] | 1.0 [0 to 2] | 2.0 [-2 to 10] | 2.0 [0 to 7] | 0.0 [-4 to 9]
  Day 56: number analyzed (Participants) | 9 | 9 | 12 | 7 | 18
  Day 56 | 1.0 [-9 to 4] | 1.0 [0 to 6] | 0.5 [-3 to 5] | 0.0 [0 to 1] | 0.0 [-3 to 12]
  Day 84: number analyzed (Participants) | 9 | 9 | 12 | 8 | 18
  Day 84 | 0.0 [-6 to 1] | 0.0 [-2 to 2] | 0.0 [-4 to 8] | 0.0 [-1 to 1] | 0.0 [-3 to 8]
Statistical Analysis 1: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.342, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 1.0, 90% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 2: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.699, Wilcoxon rank-sum test; Day 56; Median difference from baseline = 0.0, 90% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 3: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.377, Wilcoxon rank-sum test; Day 84; Median difference from baseline = -1.0, 90% CI 2-sided [-3.0 to 0.0]
Statistical Analysis 4: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.132, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 1.0, 90% CI 2-sided [0.0 to 2.0]
Statistical Analysis 5: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.292, Wilcoxon rank-sum test; Day 56; Median difference from baseline = 1.0, 90% CI 2-sided [0.0 to 2.0]
Statistical Analysis 6: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.979, Wilcoxon rank-sum test; Day 84; Median difference from baseline = 0.0, 90% CI 2-sided [-2.0 to 1.0]
Statistical Analysis 7: Comparison: LJN452 - 0.09 mg qd; Test type: Other; p = 0.102, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 2.0, 90% CI 2-sided [0.0 to 4.0]
Statistical Analysis 8: Comparison: LJN452 - 0.09 mg qd; Test type: Other; p = 0.717, Wilcoxon rank-sum test; Day 56; Median difference from baseline = 0.0, 90% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 9: Comparison: LJN452 - 0.09 mg qd; Test type: Other; p = 1.000, Wilcoxon rank-sum test; Day 84; Median difference = 0.0, 90% CI 2-sided [-2.0 to 1.0]
Statistical Analysis 10: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.142, Wilcoxon rank-sum test; Day 28; Median difference from baseline = 2.0, 90% CI 2-sided [0.0 to 5.0]
Statistical Analysis 11: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.975, Wilcoxon rank-sum test; Day 56; Median difference from baseline = 0.0, 90% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 12: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.602, Wilcoxon rank-sum test; Day 84; Median difference from baseline = 0.0, 90% CI 2-sided [-2.0 to 1.0]

13. Secondary Outcome: Change From Baseline in Global Itch Visual Analogue Scale (VAS)
Description: Baseline is defined as the latest available predose value. The Global Itch Visual Analogue Scale, a 100 mm visual analogue scale (VAS), was used to assess the severity of patients itch (ranging from 0 = none at all to 100 = the worst imaginable itch). The score range is between a minimum of 0 and a maximum of 100. The score (distance in mm from left) on the VAS was recorded by the patient marking with a line and used to test for an effect of tropifexor over placebo. The mean change from baseline in itch VAS score in each treatment group is presented.
Time Frame: Day 7, Day 14, Day 21, Day 28, Day 56, and Day 84
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: mm
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
Number analyzed (Participants) | 10 | 9 | 12 | 8 | 20
mm
  Day 7: number analyzed (Participants) | 9 | 9 | 12 | 8 | 20
  Day 7 | -2.04 [-13.84 to 9.75] | 12.08 [0.33 to 23.83] | 14.66 [4.16 to 25.16] | 27.45 [15.00 to 39.89] | 0.74 [-7.17 to 8.66]
  Day 14: number analyzed (Participants) | 9 | 9 | 12 | 7 | 20
  Day 14 | -8.04 [-19.55 to 3.48] | 13.77 [2.30 to 25.23] | 6.51 [-3.76 to 16.78] | 14.20 [1.26 to 27.13] | 6.03 [-1.70 to 13.76]
  Day 21: number analyzed (Participants) | 9 | 9 | 12 | 6 | 20
  Day 21 | 10.53 [-1.66 to 22.72] | 19.54 [7.40 to 31.68] | 7.76 [-3.11 to 18.64] | 8.65 [-5.90 to 23.20] | 2.74 [-5.44 to 10.93]
  Day 28: number analyzed (Participants) | 9 | 9 | 12 | 5 | 20
  Day 28 | 8.62 [-4.24 to 21.48] | 15.64 [2.83 to 28.44] | 1.78 [-9.69 to 13.26] | 10.50 [-5.52 to 26.51] | 1.59 [-7.04 to 10.22]
  Day 56: number analyzed (Participants) | 9 | 9 | 12 | 7 | 20
  Day 56 | -7.81 [-17.87 to 2.26] | 5.69 [-4.33 to 15.72] | -6.38 [-15.35 to 2.59] | -3.64 [-14.58 to 7.30] | 7.44 [0.68 to 14.20]
  Day 84: number analyzed (Participants) | 9 | 9 | 12 | 8 | 20
  Day 84 | -5.14 [-17.15 to 6.88] | 0.89 [-11.08 to 12.85] | -6.44 [-17.13 to 4.26] | -5.14 [-17.81 to 7.53] | 11.79 [3.73 to 19.86]
Statistical Analysis 1: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.743, ANCOVA; Day 7; Mean difference from baseline = -2.78, 90% CI 2-sided [-16.91 to 11.34], Standard Error of Mean 8.436
Statistical Analysis 2: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.093, ANCOVA; Day 14; Median difference from baseline = -14.07, 90% CI 2-sided [-27.85 to -0.28], Standard Error of Mean 8.229
Statistical Analysis 3: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.376, ANCOVA; Day 21; Median difference from baseline = 7.78, 90% CI 2-sided [-6.81 to 22.38], Standard Error of Mean 8.710
Statistical Analysis 4: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.448, ANCOVA; Day 28; Median difference from baseline = 7.03, 90% CI 2-sided [-8.36 to 22.43], Standard Error of Mean 9.187
Statistical Analysis 5: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.039, ANCOVA; Day 56; Median difference from baseline = -15.25, 90% CI 2-sided [-27.30 to -3.19], Standard Error of Mean 7.192
Statistical Analysis 6: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.054, ANCOVA; Day 84; Median difference from baseline = -16.93, 90% CI 2-sided [-31.31 to -2.54], Standard Error of Mean 8.592
Statistical Analysis 7: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.185, ANCOVA; Day 7; Median difference from baseline = 11.34, 90% CI 2-sided [-2.78 to 25.46], Standard Error of Mean 8.434
Statistical Analysis 8: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.351, ANCOVA; Day 14; Median difference from baseline = 7.74, 90% CI 2-sided [-6.05 to 21.52], Standard Error of Mean 8.226
Statistical Analysis 9: Comparison: LJN452 - 0.03 mg qd vs Placebo qd; Test type: Other; p = 0.059, ANCOVA; day 21; Median difference from baseline = 16.79, 90% CI 2-sided [2.20 to 31.38], Standard Error of Mean 8.707
Statistical Analysis 10: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.132, ANCOVA; Day 28; Median difference from baseline = 14.05, 90% CI 2-sided [-1.35 to 29.44], Standard Error of Mean 9.184
Statistical Analysis 11: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.809, ANCOVA; Day 56; Median difference from baseline = -1.75, 90% CI 2-sided [-13.80 to 10.31], Standard Error of Mean 7.190
Statistical Analysis 12: Comparison: LJN452 - 0.06 mg qd vs Placebo qd; Test type: Other; p = 0.210, ANCOVA; Day 84; Median difference from baseline = -10.90, 90% CI 2-sided [-25.29 to 3.48], Standard Error of Mean 8.590
Statistical Analysis 13: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.086, ANCOVA; day 7; Median difference from baseline = 13.92, 90% CI [0.58 to 27.25], Standard Error of Mean 7.963
Statistical Analysis 14: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.951, ANCOVA; Day 14; Median difference from baseline = 0.48, 90% CI 2-sided [-12.57 to 13.53], Standard Error of Mean 7.787
Statistical Analysis 15: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.545, ANCOVA; day 21; Median difference from baseline = 5.02, 90% CI 2-sided [-8.79 to 18.83], Standard Error of Mean 8.244
Statistical Analysis 16: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.982, ANCOVA; Day 28; Median difference from baseline = 0.19, 90% CI 2-sided [-14.38 to 14.77], Standard Error of Mean 8.697
Statistical Analysis 17: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.047, ANCOVA; day 56; Median difference from baseline = -13.82, 90% CI 2-sided [-25.21 to -2.43], Standard Error of Mean 6.797
Statistical Analysis 18: Comparison: LJN452 - 0.09 mg qd vs Placebo qd; Test type: Other; p = 0.029, ANCOVA; Day 84; Median difference from baseline = -18.23, 90% CI 2-sided [-31.81 to -4.64], Standard Error of Mean 8.110
Statistical Analysis 19: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.004, ANCOVA; Day 7; Median difference from baseline = 26.70, 90% CI 2-sided [11.97 to 41.44], Standard Error of Mean 8.799
Statistical Analysis 20: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.370, ANCOVA; Day 14; Median difference from baseline = 8.17, 90% CI 2-sided [-6.96 to 23.29], Standard Error of Mean 9.032
Statistical Analysis 21: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.558, ANCOVA; Day 21; Median difference from baseline = 5.90, 90% CI 2-sided [-10.86 to 22.66], Standard Error of Mean 10.014
Statistical Analysis 22: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.418, ANCOVA; Day 28; Median difference from baseline = 8.91, 90% CI 2-sided [-9.34 to 27.15], Standard Error of Mean 10.911
Statistical Analysis 23: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.156, ANCOVA; Day 56; Median difference from baseline = -11.08, 90% CI 2-sided [-23.95 to 1.80], Standard Error of Mean 7.690
Statistical Analysis 24: Comparison: LJN452 - 0.15 mg qd vs Placebo qd; Test type: Other; p = 0.064, ANCOVA; Day 84; Median difference from baseline = -16.93, 90% CI 2-sided [-31.94 to -1.92], Standard Error of Mean 8.961

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 56 days post last dose.
Arm/Group | LJN452 - 0.03 mg qd | LJN452 - 0.06 mg qd | LJN452 - 0.09 mg qd | LJN452 - 0.15 mg qd | Placebo qd
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/12 | 0/8 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/12 | 0/8 | 0/21
Other Adverse Events (participants affected / at risk) | 9/11 | 8/9 | 11/12 | 8/8 | 16/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LJN452 - 0.03 mg qd (N=11) | LJN452 - 0.06 mg qd (N=9) | LJN452 - 0.09 mg qd (N=12) | LJN452 - 0.15 mg qd (N=8) | Placebo qd (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Trifascicular block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 3
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 1
Overgrowth bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6 | 5 | 7 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02516605/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT02516605/SAP_001.pdf